CLINICAL TRIAL: NCT02647736
Title: Kinetics of Copeptin in Healthy Volunteers - a Prospective International Study
Brief Title: Copeptin in Normal- to Hyperosmolar States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Mirjam Christ-Crain, Prof. Dr. med., University Hospital, Basel, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CoNorm
Record Dates: First submitted 2015-12-23; First posted 2016-01-06 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Copeptin Blood Values

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Copeptin values in normo- to hyperosmolar states (Experimental)
  Interventions: Other: Hypertonic saline infusion

INTERVENTIONS:
Other: Hypertonic saline infusion

SUMMARY:
Kinetics of Copeptin in response to osmotic alterations in healthy volunteers

DETAILED DESCRIPTION:
Construction of the standard area of copeptin release in the normo- and hyperosmolar state and its half-life based on ist decline during hypoosmotic Suppression in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age 18
* no severe comorbidities
* no medication (except contraceptives)
* baseline sodium Level 135-145mmol/l
* euvolemic status

Exclusion Criteria:

* history of heart failure
* liver cirrhosis
* kidney disease (GFR <60ml/min)
* anemia
* uncontrolled Hypertension
* pregnancy
* Diabetes mellitus
* BMI >28kg/m2
* other severe disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physiological relationship between Serum osmolality and Plasma copeptin release. | beginning and end of protocol, up to 8 hours
  Copeptin and Blood osmolality will be measured concomitantly while hypertonic saline is infused. The infusion is continued until a hyperosmolar state is reached (defined with a sodium-level of 150mmol/l).
  Definition of an area of normality describing the physiological relationship between Serum osmolality and Plasma copeptin release in normo- to hyperosmolar states.
Half life of Copeptin | beginning and end of protocol, up to 8 hours
  Calculation of Copeptin half-life based on its decline during hypoosmotic suppression (oral waterload and glucose 5%-infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- University Hospital Würzburg, Würzburg, Germany
- University hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Sailer CO, Refardt J, Blum CA, Schnyder I, Molina-Tijeras JA, Fenske W, Christ-Crain M. Validity of different copeptin assays in the differential diagnosis of the polyuria-polydipsia syndrome. Sci Rep. 2021 May 12;11(1):10104. doi: 10.1038/s41598-021-89505-9. PMID 33980941
- [Derived] Fenske WK, Schnyder I, Koch G, Walti C, Pfister M, Kopp P, Fassnacht M, Strauss K, Christ-Crain M. Release and Decay Kinetics of Copeptin vs AVP in Response to Osmotic Alterations in Healthy Volunteers. J Clin Endocrinol Metab. 2018 Feb 1;103(2):505-513. doi: 10.1210/jc.2017-01891. PMID 29267966